CLINICAL TRIAL: NCT04997733
Title: Fecal Microbiota Transplantation in Crohn's Disease as Relay After Anti-TNF Withdrawal
Acronym: MIRACLE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CRB-HUEP (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP190183; 2019-003816-29 (EudraCT Number)
Record Dates: First submitted 2021-07-05; First posted 2021-08-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Crohn Disease
Keywords: Crohn disease; Inflammatory bowel disease; Fecal microbiota transplantation
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal microbiota (Experimental): Patients receiving the fecal microbiota transplantation (FMT) in 3 times after inclusion and randomisation (endoscopic and oral)
  Interventions: Drug: Fecal Microbiota Transplantation (FMT)
- Sham-transplantation (Sham Comparator): Patients receiving the sham-transplantation in 3 times after inclusion and randomisation (endoscopic and oral)
  Interventions: Drug: Sham-transplantation (placebo)

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation (FMT) — The colonoscopy for FMT will be planned between 7 and 14 days after the last adalimumab or sub-cutaneous infliximab administration and 6 weeks +/- 7 days after the last intravenous infliximab administration 14 and 28 days following the last sub-cutaneous golimumab administration. After colon cleansing using polyethylene glycol, the patient will have a colonoscopy under general anesthesia. The patient will then receive either FMT (frozen preparation of 50g of stools in 300ml of saline (NaCl 0.9%), (FMT vehicle in the terminal ileum or the colon.
  At W12 and W24 after first colonoscopy, the patient receives treatment by capsule (15 capsules contain 0.8g of stools by visit).
  Arms: Fecal microbiota
Drug: Sham-transplantation (placebo) — The colonoscopy for sham-transplantation will be planned between 7 and 14 days after the last adalimumab or sub-cutaneous infliximab administration and 6 weeks +/- 7 days after the last intravenous infliximab administration, 14 and 28 days following the last sub-cutaneous golimumab administration. After colon cleansing using polyethylene glycol, the patient will have a colonoscopy under general anesthesia. The patient will then receive either sham transplantation (frozen preparation of NaCl 0.9% with 10% glycerol) in the terminal ileum or the colon.
  At S12 and S24 after first colonoscopy, the patient receives treatment by capsule (15 capsules contain placebo).
  Arms: Sham-transplantation

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory bowel disease. CD pathogenesis remains poorly understood but involves an inappropriate immune response toward an unbalanced gut microbiota in predisposed hosts.

The purpose of this study is to evaluate de clinical efficacy of the fecal microbiota transplantation (FMT) as a maintenance treatment following anti-TNF agent withdrawal in CD's patient.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic inflammatory bowel disease affecting approximately 120000 patients in France, mostly at young age, and altering their quality of life.

Immunosuppressive treatments in CD are expensive and associated with potentially severe complications.

Alternative treatment strategies are thus required. This is particularly the case for CD patients in remission under anti-TNF agents for which no specific recommendation are available.

CD pathogenesis remains poorly understood but involves an inappropriate immune response toward an unbalanced gut microbiota in predisposed hosts.

Fecal microbiota transplantation (FMT) is currently recommended for treating recurrent Clostridium difficile infection. Although the pathogenesis involved in CD differs, FMT is a potential therapeutic strategy that could restore the appropriate host-microbiota crosstalk by transferring a healthy microbiota in a CD patient. However, as the gut microbiota is dramatically altered by intestinal inflammation, transferring a massive amount of microbes in an inflamed gut with epithelial barrier disruption might be a suboptimal strategy and could even have detrimental effects by allowing bacterial translocation.

Results of randomized controlled trial (RCT) in CD are lacking to date. We performed a pilot RCT (NCT02097797), evaluating the impact of a single FMT in 18 CD patients who achieved remission by corticosteroid treatment. A higher rate of steroid free clinical remission was observed in the FMT arm at 24 weeks (57.1% vs 33.3% in FMT and control arm respectively). CD Endoscopic Index of Severity was also improved at 6 weeks in FMT (median 8.5 vs 3.5 p=0.03) but not in sham group (median 2.4 vs 2.7 p=0.8). Moreover, the only 2 patients who early relapsed in the FMT group were those who did not show any engraftment of donor microbiota at week 6. These promising data, currently submitted for publication, suggest that using FMT as a maintenance treatment in CD can be effective. However, these promising findings need to be confirmed by a Phase III RCT.

ELIGIBILITY:
Inclusion Criteria for patients :

* Age ≥ 18 years and < 75 years
* Crohn's disease (according to the Lennard-Jones criteria) for at least 6 months
* Patient in steroid-free clinical remission for at least 6 months under anti-TNF agent (no clinical evidence of flare nor change in Crohn's disease specific treatment (anti-TNF, immunosuppressive, …) within 6 months before inclusion) and CDAI <150 the week before inclusion) and willing to withdraw anti-TNF treatment
* Female of child-bearing age with an active contraception and this during at least the period of treatment (week 52)
* Patient with health insurance
* Informed Written consent

Inclusion Criteria for healthy volunteer donor :

* Age ≥ 18 years and < 50 years
* 17 kg/m² < body mass index < 30 kg/m²
* Regular bowel movement defined as at least 1 stool every other day and maximum 2 stools per day
* Subject with health insurance (AME excepted)
* Informed written consent

Exclusion Criteria for patients :

* Crohn's Disease complication requiring surgical treatment
* Contraindication to colonoscopy or anesthesia
* Pregnancy or breastfeeding during the study (Cf. Addendum 4)
* Diagnosis of Crohn's disease restricted to the upper gastrointestinal tract (oesophagus, stomach, duodenum, jejunum)
* Patient with active perineal disease (defined as evidence of perineal abscess or active draining fistula or presence of seton or presence of perineal ulceration)
* History of more than one small bowel resection or small intestine resection > 1 meter
* Current stoma (Ileostomy or a colostomy) or stoma in the last 6 months or any other intra-abdominal surgery within 3 months prior to inclusion
* Participation in any other interventional study
* Patient under legal protection

Exclusion Criteria for healthy volunteer donor :

- For details, please see protocol

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2027-05-22 (Estimated); Study Completion 2029-07-22 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical efficacy of FMT versus sham transplantation as a maintenance treatment following anti-TNF agent withdrawal in patients with Crohn's disease in steroid-free clinical remission for at least 6 months under anti-TNF agent | 52 weeks after FMT or sham-transplantation
  Clinical remission (defined by a Crohn's disease activity index (CDAI) <150) at week 52 (V8) without any flare between week 0 (colonoscopy (V2)) and week 52 (V8). Flare is defined by a CDAI (Addendum 2) above 250 or between 150 points and 250 points with a 70-point increase from baseline over 2 consecutive weeks and the need

SECONDARY OUTCOMES:
Relapse free survival | 52 weeks after FMT or sham-transplantation
  Relapse free survival rate from week 0 (V2) to week 52 (V8)

OTHER OUTCOMES:
Mucosal healing | 52 weeks after FMT or sham-transplantation
  Proportion of endoscopic remission (SES-CD ≤2) at week 52 (V8) and change (in %) in endoscopic score (SES-CD) between week 0 (V2) and 52 (V8)
Clinical remission | 52 weeks after FMT or sham-transplantation
  Clinical remission defined by a CDAI < 150 at week 52
Endoscopic remission | 52 weeks after FMT or sham-transplantation
  Endoscopic remission defined by a SES-CD ≤ 2 at week 52
Changes in inflammation 1 | 6, 12, 24, 36, 48 and 52 weeks after TMF or sham-transplantation
  Measures of inflammation: blood cell count
Changes in inflammation 2 | 6, 12, 24, 36, 48 and 52 weeks after TMF or sham-transplantation
  Measures of inflammation: C reactive protein (CRP) level
Changes in inflammation 3 | 6, 12, 24, 36, 48 and 52 weeks after TMF or sham-transplantation
  Measures of inflammation: fecal calprotectin
Changes in intestinal microbiota composition | 6, 12, 24, 36, 48 and 52 weeks after TMF or sham-transplantation
  Microbiota composition and diversity using 16s sequencing technology

CONTACTS AND LOCATIONS:
Overall Officials: Harry SOKOL, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Gastroenterology Department of Saint Antoine Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ananthakrishnan AN. Epidemiology and risk factors for IBD. Nat Rev Gastroenterol Hepatol. 2015 Apr;12(4):205-17. doi: 10.1038/nrgastro.2015.34. Epub 2015 Mar 3. PMID 25732745
- [Background] Angelberger S, Reinisch W, Makristathis A, Lichtenberger C, Dejaco C, Papay P, Novacek G, Trauner M, Loy A, Berry D. Temporal bacterial community dynamics vary among ulcerative colitis patients after fecal microbiota transplantation. Am J Gastroenterol. 2013 Oct;108(10):1620-30. doi: 10.1038/ajg.2013.257. Epub 2013 Sep 24. PMID 24060759
- [Background] Beaugerie L, Itzkowitz SH. Cancers Complicating Inflammatory Bowel Disease. N Engl J Med. 2015 Jul 9;373(2):195. doi: 10.1056/NEJMc1505689. No abstract available. PMID 26154801
- [Background] Ben-Horin S, Chowers Y. Review article: loss of response to anti-TNF treatments in Crohn's disease. Aliment Pharmacol Ther. 2011 May;33(9):987-95. doi: 10.1111/j.1365-2036.2011.04612.x. Epub 2011 Mar 2. PMID 21366636
- [Background] Best WR, Becktel JM, Singleton JW, Kern F Jr. Development of a Crohn's disease activity index. National Cooperative Crohn's Disease Study. Gastroenterology. 1976 Mar;70(3):439-44. PMID 1248701
- [Background] Borody T, Fischer M, Mitchell S, Campbell J. Fecal microbiota transplantation in gastrointestinal disease: 2015 update and the road ahead. Expert Rev Gastroenterol Hepatol. 2015;9(11):1379-91. doi: 10.1586/17474124.2015.1086267. Epub 2015 Sep 28. PMID 26414076
- [Background] Colman RJ, Rubin DT. Fecal microbiota transplantation as therapy for inflammatory bowel disease: a systematic review and meta-analysis. J Crohns Colitis. 2014 Dec;8(12):1569-81. doi: 10.1016/j.crohns.2014.08.006. Epub 2014 Sep 13. PMID 25223604
- [Background] Cui B, Li P, Xu L, Zhao Y, Wang H, Peng Z, Xu H, Xiang J, He Z, Zhang T, Nie Y, Wu K, Fan D, Ji G, Zhang F. Step-up fecal microbiota transplantation strategy: a pilot study for steroid-dependent ulcerative colitis. J Transl Med. 2015 Sep 12;13:298. doi: 10.1186/s12967-015-0646-2. PMID 26363929
- [Background] Cui B, Feng Q, Wang H, Wang M, Peng Z, Li P, Huang G, Liu Z, Wu P, Fan Z, Ji G, Wang X, Wu K, Fan D, Zhang F. Fecal microbiota transplantation through mid-gut for refractory Crohn's disease: safety, feasibility, and efficacy trial results. J Gastroenterol Hepatol. 2015 Jan;30(1):51-8. doi: 10.1111/jgh.12727. PMID 25168749
- [Background] D'Haens G, Sandborn WJ, Feagan BG, Geboes K, Hanauer SB, Irvine EJ, Lemann M, Marteau P, Rutgeerts P, Scholmerich J, Sutherland LR. A review of activity indices and efficacy end points for clinical trials of medical therapy in adults with ulcerative colitis. Gastroenterology. 2007 Feb;132(2):763-86. doi: 10.1053/j.gastro.2006.12.038. Epub 2006 Dec 20. No abstract available. PMID 17258735
- [Background] Debast SB, Bauer MP, Kuijper EJ; European Society of Clinical Microbiology and Infectious Diseases. European Society of Clinical Microbiology and Infectious Diseases: update of the treatment guidance document for Clostridium difficile infection. Clin Microbiol Infect. 2014 Mar;20 Suppl 2:1-26. doi: 10.1111/1469-0691.12418. PMID 24118601
- [Background] Grinspan AM, Kelly CR. Fecal Microbiota Transplantation for Ulcerative Colitis: Not Just Yet. Gastroenterology. 2015 Jul;149(1):15-8. doi: 10.1053/j.gastro.2015.05.030. Epub 2015 May 27. No abstract available. PMID 26021232
- [Background] Kennedy NA, Warner B, Johnston EL, Flanders L, Hendy P, Ding NS, Harris R, Fadra AS, Basquill C, Lamb CA, Cameron FL, Murray CD, Parkes M, Gooding I, Ahmad T, Gaya DR, Mann S, Lindsay JO, Gordon J, Satsangi J, Hart A, McCartney S, Irving P; UK Anti-TNF withdrawal study group; Lees CW. Relapse after withdrawal from anti-TNF therapy for inflammatory bowel disease: an observational study, plus systematic review and meta-analysis. Aliment Pharmacol Ther. 2016 Apr;43(8):910-923. doi: 10.1111/apt.13547. Epub 2016 Feb 19. PMID 26892328
- [Background] Kelly CR, Ihunnah C, Fischer M, Khoruts A, Surawicz C, Afzali A, Aroniadis O, Barto A, Borody T, Giovanelli A, Gordon S, Gluck M, Hohmann EL, Kao D, Kao JY, McQuillen DP, Mellow M, Rank KM, Rao K, Ray A, Schwartz MA, Singh N, Stollman N, Suskind DL, Vindigni SM, Youngster I, Brandt L. Fecal microbiota transplant for treatment of Clostridium difficile infection in immunocompromised patients. Am J Gastroenterol. 2014 Jul;109(7):1065-71. doi: 10.1038/ajg.2014.133. Epub 2014 Jun 3. PMID 24890442
- [Background] Kelly CR, Kahn S, Kashyap P, Laine L, Rubin D, Atreja A, Moore T, Wu G. Update on Fecal Microbiota Transplantation 2015: Indications, Methodologies, Mechanisms, and Outlook. Gastroenterology. 2015 Jul;149(1):223-37. doi: 10.1053/j.gastro.2015.05.008. Epub 2015 May 15. PMID 25982290
- [Background] Khor B, Gardet A, Xavier RJ. Genetics and pathogenesis of inflammatory bowel disease. Nature. 2011 Jun 15;474(7351):307-17. doi: 10.1038/nature10209. PMID 21677747
- [Background] Lamas B, Richard ML, Leducq V, Pham HP, Michel ML, Da Costa G, Bridonneau C, Jegou S, Hoffmann TW, Natividad JM, Brot L, Taleb S, Couturier-Maillard A, Nion-Larmurier I, Merabtene F, Seksik P, Bourrier A, Cosnes J, Ryffel B, Beaugerie L, Launay JM, Langella P, Xavier RJ, Sokol H. CARD9 impacts colitis by altering gut microbiota metabolism of tryptophan into aryl hydrocarbon receptor ligands. Nat Med. 2016 Jun;22(6):598-605. doi: 10.1038/nm.4102. Epub 2016 May 9. PMID 27158904
- [Background] Le Chatelier E, Nielsen T, Qin J, Prifti E, Hildebrand F, Falony G, Almeida M, Arumugam M, Batto JM, Kennedy S, Leonard P, Li J, Burgdorf K, Grarup N, Jorgensen T, Brandslund I, Nielsen HB, Juncker AS, Bertalan M, Levenez F, Pons N, Rasmussen S, Sunagawa S, Tap J, Tims S, Zoetendal EG, Brunak S, Clement K, Dore J, Kleerebezem M, Kristiansen K, Renault P, Sicheritz-Ponten T, de Vos WM, Zucker JD, Raes J, Hansen T; MetaHIT consortium; Bork P, Wang J, Ehrlich SD, Pedersen O. Richness of human gut microbiome correlates with metabolic markers. Nature. 2013 Aug 29;500(7464):541-6. doi: 10.1038/nature12506. PMID 23985870
- [Background] Lee CH, Steiner T, Petrof EO, Smieja M, Roscoe D, Nematallah A, Weese JS, Collins S, Moayyedi P, Crowther M, Ropeleski MJ, Jayaratne P, Higgins D, Li Y, Rau NV, Kim PT. Frozen vs Fresh Fecal Microbiota Transplantation and Clinical Resolution of Diarrhea in Patients With Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2016 Jan 12;315(2):142-9. doi: 10.1001/jama.2015.18098. PMID 26757463
- [Background] Lennard-Jones JE. Classification of inflammatory bowel disease. Scand J Gastroenterol Suppl. 1989;170:2-6; discussion 16-9. doi: 10.3109/00365528909091339. PMID 2617184
- [Background] Manichanh C, Borruel N, Casellas F, Guarner F. The gut microbiota in IBD. Nat Rev Gastroenterol Hepatol. 2012 Oct;9(10):599-608. doi: 10.1038/nrgastro.2012.152. Epub 2012 Aug 21. PMID 22907164
- [Background] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Background] Paramsothy S, Kamm MA, Kaakoush NO, Walsh AJ, van den Bogaerde J, Samuel D, Leong RWL, Connor S, Ng W, Paramsothy R, Xuan W, Lin E, Mitchell HM, Borody TJ. Multidonor intensive faecal microbiota transplantation for active ulcerative colitis: a randomised placebo-controlled trial. Lancet. 2017 Mar 25;389(10075):1218-1228. doi: 10.1016/S0140-6736(17)30182-4. Epub 2017 Feb 15. PMID 28214091
- [Background] Rossen NG, Fuentes S, van der Spek MJ, Tijssen JG, Hartman JH, Duflou A, Lowenberg M, van den Brink GR, Mathus-Vliegen EM, de Vos WM, Zoetendal EG, D'Haens GR, Ponsioen CY. Findings From a Randomized Controlled Trial of Fecal Transplantation for Patients With Ulcerative Colitis. Gastroenterology. 2015 Jul;149(1):110-118.e4. doi: 10.1053/j.gastro.2015.03.045. Epub 2015 Mar 30. PMID 25836986
- [Background] Sokol H, Leducq V, Aschard H, Pham HP, Jegou S, Landman C, Cohen D, Liguori G, Bourrier A, Nion-Larmurier I, Cosnes J, Seksik P, Langella P, Skurnik D, Richard ML, Beaugerie L. Fungal microbiota dysbiosis in IBD. Gut. 2017 Jun;66(6):1039-1048. doi: 10.1136/gutjnl-2015-310746. Epub 2016 Feb 3. PMID 26843508
- [Background] Sokol H, Galperine T, Kapel N, Bourlioux P, Seksik P, Barbut F, Scanzi J, Chast F, Batista R, Joly F, Joly AC, Collignon A, Guery B, Beaugerie L; French Group of Faecal microbiota Transplantation (FGFT). Faecal microbiota transplantation in recurrent Clostridium difficile infection: Recommendations from the French Group of Faecal microbiota Transplantation. Dig Liver Dis. 2016 Mar;48(3):242-7. doi: 10.1016/j.dld.2015.08.017. Epub 2015 Sep 7. PMID 26433619
- [Background] Sokol H. Toward Rational Donor Selection in Faecal Microbiota Transplantation for IBD. J Crohns Colitis. 2016 Apr;10(4):375-6. doi: 10.1093/ecco-jcc/jjw005. Epub 2016 Jan 7. No abstract available. PMID 26746170
- [Background] Sokol H, Lalande V, Landman C, Bourrier A, Nion-Larmurier I, Rajca S, Kirchgesner J, Seksik P, Cosnes J, Barbut F, Beaugerie L. Clostridium difficile infection in acute flares of inflammatory bowel disease: A prospective study. Dig Liver Dis. 2017 Jun;49(6):643-646. doi: 10.1016/j.dld.2017.01.162. Epub 2017 Jan 30. PMID 28215602
- [Background] Suskind DL, Singh N, Nielson H, Wahbeh G. Fecal microbial transplant via nasogastric tube for active pediatric ulcerative colitis. J Pediatr Gastroenterol Nutr. 2015 Jan;60(1):27-9. doi: 10.1097/MPG.0000000000000544. PMID 25162366
- [Background] Toruner M, Loftus EV Jr, Harmsen WS, Zinsmeister AR, Orenstein R, Sandborn WJ, Colombel JF, Egan LJ. Risk factors for opportunistic infections in patients with inflammatory bowel disease. Gastroenterology. 2008 Apr;134(4):929-36. doi: 10.1053/j.gastro.2008.01.012. Epub 2008 Jan 11. PMID 18294633
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Vermeire S, Joossens M, Verbeke K, Wang J, Machiels K, Sabino J, Ferrante M, Van Assche G, Rutgeerts P, Raes J. Donor Species Richness Determines Faecal Microbiota Transplantation Success in Inflammatory Bowel Disease. J Crohns Colitis. 2016 Apr;10(4):387-94. doi: 10.1093/ecco-jcc/jjv203. Epub 2015 Oct 29. PMID 26519463
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514
- [Background] Youngster I, Mahabamunuge J, Systrom HK, Sauk J, Khalili H, Levin J, Kaplan JL, Hohmann EL. Oral, frozen fecal microbiota transplant (FMT) capsules for recurrent Clostridium difficile infection. BMC Med. 2016 Sep 9;14(1):134. doi: 10.1186/s12916-016-0680-9. PMID 27609178
- See also: Related Info — https://research.monash.edu/en/publications/short-duration-low-intensity-pooled-faecal-microbiota-transplanta